CLINICAL TRIAL: NCT06648759
Title: The Role of a Vagal Stimulator to Reduce the Frequency and Duration on Nasogastric Tube Following Abdominal Surgery
Brief Title: Vagal Stimulator to Reduce Nasogastric Tube Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jacques E. Chelly (Other)
Responsible Party: Sponsor-Investigator, Jacques E. Chelly, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY24070152
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Nasogastric Tube Intubation

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects will be 2:1 randomized to the Vagal Nerve Stimulator Group or the Placebo Group, respectively.
  A blinded study team member will use a standard, active device to establish the threshold of current required to stimulate the vagal nerve via an electrode placed on each side of the neck. The study device will be placed after surgery once an NG tube has been administered. This study device placement and adjustment may happen anywhere from the PACU to the hospital ward level, dependent on the NG tube placement timing, but it will be done in a private setting for confidential safeguards.
  According to the standard operative procedure of the vagal stimulator, this current threshold is achieved by (1) increasing the current until the patient feels the sensation, and then (2) reducing the current until the patient no longer feels the current. When this is established, a research-specific device (either active or sham, based on the randomization assignment) will be connected to the elect
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vagal Nerve Stimulator Group (Experimental): This arm of the study will be randomly assigned to receive the active vagal nerve stimulator device which is placed via electrodes on each side of the neck. The active device will experience two 45-minute sessions daily of vagal nerve stimulation until their Nasogastric (NG) tube is removed.
  Interventions: Device: Vagal Nerve Stimulator
- Placebo Vagal Nerve Stimulator Group (Sham Comparator): This arm of the study will be randomly assigned to receive a sham device that mirrors that of the active vagal nerve stimulator devices. The sham device arm will experience two 45-minute sessions daily of placebo vagal nerve stimulation until their Nasogastric (NG) tube is removed.
  Interventions: Device: Placebo Vagal Nerve Stimulator

INTERVENTIONS:
Device: Vagal Nerve Stimulator — The vagal nerve stimulator device is a nonsignificant risk device that provides electrical impulses to the vagus nerve, located in the neck and ear regions. The device (pulse generator) and a wire lead (insulated wire) with electrodes on the end of the wire will send the electrical signals along the vagus nerve to your brainstem to activate various neurochemical coordinates.
  Arms: Vagal Nerve Stimulator Group
Device: Placebo Vagal Nerve Stimulator — The sham vagal nerve stimulator device is a nonsignificant risk device that mirrors that of the active stimulator but does not provide electrical impulses to the vagus nerve.
  Arms: Placebo Vagal Nerve Stimulator Group

SUMMARY:
Abdominal surgery, laparoscopic or open, is frequently performed at UPMC Shadyside hospital. One of the most frequent complications following abdominal surgery is a postoperative ileus. Although postoperative ileus may be the result of obstruction or leakage, in most cases postoperative ileus (POI) is the result of local irritation because of fluid overload, exogenous opioids, neurohormonal dysfunction, gastrointestinal stretch, local bleeding and inflammation. POI usually lasts between 2 to 7 days. In most cases, a nasogastric tube (NG tube) is used to relieve that gastric pressure until the resolution of the POI. The placement of a NG tube can lead to a local trauma, bleeding and pain. Pain represents a major complaint among those with POI, often contributing to prolonged hospital stays.

DETAILED DESCRIPTION:
Abdominal surgery, laparoscopic or open, is frequently performed at UPMC Shadyside hospital. One of the most frequent complications following abdominal surgery is a postoperative ileus. Although postoperative ileus may be the result of obstruction or leakage, in most cases postoperative ileus (POI) is the result of local irritation because of fluid overload, exogenous opioids, neurohormonal dysfunction, gastrointestinal stretch, local bleeding and inflammation. POI usually lasts between 2 to 7 days. In most cases, a nasogastric tube (NG tube) is used to relieve that gastric pressure until the resolution of the POI. The placement of a NG tune can lead to a local trauma, bleeding and pain. Pain represents a major complaint among those with POI, often contributing to prolonged hospital stays.

It has been well established that bile function is modulated by the vagal nerve. Therefore, a non-invasive vagal stimulation administered post-operatively may facilitate the resolution of POI, accelerate the return to bile function and shorter the hospital length of stay following major abdominal surgery. Anecdotally, the use of a vagal nerve stimulator has been shown to avoid the placement of a NG tube.

In most cases, postoperative ileus is considered a benign and reversible complication that occurs in 10-30% of patients following abdominal surgery. The use of anesthesia, the use of opioids and anti-inflammatory drugs, hypokalemia, local inflammation, local hematoma, can all contribute to the development of a POI, and its treatment often requires the placement of a NG tube. The placement of a NG tube is not always effective if it is not positioned properly and is associated of a local trauma, misplacement of the NG tube, prolonged pain, and hospital stay. It is always very uncomfortable for the patient. Since the gastro-intestinal motility is regulated by the vagal nerve, the use of non-invasive vagal nerve stimulator may represent an interesting technique to reduce the frequency of this complications associated with the use of a nasogastric tube including local trauma, misplacement and pain on insertion, and constant pain as long as the NG tube remain in place.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 and older) undergoing laparoscopic or open colorectal surgery, or any major abdominal surgeries at UPMC Shadyside
* Development of post-operative ileus
* Anticipation of a nasogastric (ng) tube being placed

Exclusion Criteria:

* Pregnant subjects
* Subjects who are unable to read, write, or speak English fluently
* Subjects who have a developmental or neurological disorder and are not cognitively able to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Duration of use of nasogastric (NG) tube | Up to 30 days following surgery
  The duration of use of nasogastric (NG) tube will be reported as total of minutes the NG tube is placed and reported in each group as mean(SD) in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques E Chelly, MD, PhD, MBA, Principal Investigator — University of Pittsburgh, UPMC
Locations (1):
- UPMC Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No